CLINICAL TRIAL: NCT07018011
Title: Comparison of Conventional Versus Transverse Mini-Incision Technique for Carpal Tunnel Release: A Randomized Controlled Trial
Brief Title: Comparison of Conventional Versus Transverse Mini-Incision Technique for Carpal Tunnel Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRKASHIFSAHIWAL
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional open CTR (Experimental): Conventional open CTR involved making a longitudinal incision in the wrist, typically along the median palmar crease, to access and release the transverse carpal ligament.
  Interventions: Procedure: Conventional open CTR
- Transverse mini-incision technique (Experimental): Mini-incision CTR involved a smaller incision than traditional CTR procedures, aiming to minimize scarring and improve recovery time.
  Interventions: Procedure: Transverse mini-incision technique

INTERVENTIONS:
Procedure: Conventional open CTR — Conventional open CTR involved making a longitudinal incision in the wrist, typically along the median palmar crease, to access and release the transverse carpal ligament.
  Arms: Conventional open CTR
Procedure: Transverse mini-incision technique — Mini-incision CTR involved a smaller incision than traditional CTR procedures, aiming to minimize scarring and improve recovery time.
  Arms: Transverse mini-incision technique

SUMMARY:
This study aimed at to fill the gaps by comparing the surgical outcomes of the conventional versus transverse mini-incision technique for carpal tunnel syndrome in terms of pain and functional outcomes.

DETAILED DESCRIPTION:
The study findings would be helpful in determining the superiority of one surgical technique over the other for carpal tunnel release so that a quicker return to normal activities and work for those patients could be achieved, causing less pain and scarring. Due to frequent healthcare visits, quality of life can also be improved along with a decrease in morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Any genders
* Aged between 18 and 70 years
* Presenting with symptoms of carpal tunnel syndrome for at least 3 months duration, and having a VAS score > 4.

Exclusion Criteria:

* Patients with wrists with thenar atrophy
* Those who had previous CTR surgery
* Local injection for CTS
* Pregnant females
* Patients suffering from inflammatory arthropathy
* Polyneuropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Pain severity | 9 months
  A score percentage of 0-40 on the visual analog scale was graded as good, 50-60 as fair, and 70-100 as poor
Functional outcome | 9 months
  On functional severity scale, a score percentage of 20-45% was graded as good, 46-60% was graded as fair, and 61-100% was graded as poor.

CONTACTS AND LOCATIONS:
Overall Officials: Kashif Raza, FCPS, Principal Investigator — Sahiwal Teaching Hospital, Sahiwal; Muhammad Rashid, FCPS, Study Director — Sahiwal Teaching Hospital, Sahiwal
Locations (1):
- Sahiwal Teaching Hospital, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.